CLINICAL TRIAL: NCT06528366
Title: High Definition Transcranial Continuous Current Stimulation and Consumption of Chlorella Pyrenoidosa as Adjuvant Treatment for Heart Failure With Reduced Ejection Fraction
Brief Title: Heart Failure With Reduced Ejection Fraction: Adjuvant Therapy With Neurostimulation and Chlorella Pyrenoidosa (HD-tDCS)
Acronym: HD-tDCS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Collaborators: The City College of New York (Other)
Responsible Party: Principal Investigator, Suellen Andrade, PhD Suellen Marinho Andrade, Federal University of Paraíba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HD-tDCS/Chlorella p./HFREF
Record Dates: First submitted 2024-07-21; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure, Reduced Ejection Fraction; Vitamin B12 Deficiency
Keywords: High-density Transcranial Direct Current Stimulation; Vitamin B12 Deficiency; Heart Failure with Reduced Ejection Fraction; Functional Food; Chlorella pyrenoidosa
MeSH Terms: conditions — Heart Failure, Systolic; Vitamin B 12 Deficiency

STUDY DESIGN:
Intervention Model Description: Crossover Study Experimental Group Hospital phase (Group 1): Patients will receive 3mA current for 20 minutes with anodal stimulation through HD-tDCS (4x1) with 5 sessions on 5 consecutive days and before the surgical procedure.
  Control Group (2) Sham: Patients receive the simulated HD-tDCS anodic current (4x1) with 3mA that accelerates for 30 seconds and decelerates for another 30 seconds, 5 sessions on 5 consecutive days and before the surgical procedure .
  Washout period - surgery and recovery for discharge (on average 15 days). Experimental Group Outpatient phase (Group 1) - active for Chlorella pyrenoidosa - consume 10 tablets per day of Chlorella p for 30 days. (5g/day) and must return within 30 days for evaluation.
  Control Group 2 - will not consumption of Chlorella pyrenoidosa and must return within 30 days for evaluation.
Who Masked: Participant, Care Provider
Masking Description: The research includes the responsible researcher, assistant and collaborator. The Collaborating Researcher is responsible for applying the technique to the patient not knowing which stimulus will be true or sham. He must apply the research tools and fill out de forms. The Collaborating Researcher should alert the Main Researcher and Assistant Research if regards signs or symptoms in patient resulting adverse effects.
  In this way, the patient and the Collaborating Researcher are blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group HD-tDCS (Hospital fase) (Experimental): Experimental group HD-tDCS will be started at hospital fase when the patients will be randomly enrolled into tis group. They will receive 3mA current for 20 minutes with anodal stimulation through HD-tDCS (4x1) to the left dorsolateral prefrontal cortex, with 5 sessions on 5 consecutive days and before the surgical procedure.
  Interventions: Device: High Definition Transcranial Direct Current Stimulation
- Sham Group (Hospital Fase) (Sham Comparator): Sham Group (Hospital Fase) will be started at hospital fase when the patients will be randomly enrolled into tis group. They will receive simulated HD-tDCS anodic current (4x1) to the left dorsolateral prefrontal cortex with 3mA that accelerates for 30 seconds and decelerates for another 30 seconds, 5 sessions on 5 consecutive days and before the surgical procedure.
  Interventions: Device: High Definition Transcranial Direct Current Stimulation
- Experimental Group Chlorella pyrenoidosa (Outpatient phase) (Active Comparator): The groups are inverted due to the crossover design, so the previous sham group becomes the active group for Chlorella p consumption after the washout . So, this group must consume 10 tablets per day of Chlorella p for 30 days. (5g/day) and must return within 30 days for evaluation.
  Interventions: Dietary Supplement: Chlorella pyrenoidosa
- Control Group (Outpatient phase) (No Intervention): This group was inverted using the crossover method, so the active group for HD-tDCS in the previous phase and after the washout is inverted and becomes the control group in this phase. So, they will not receive intervention and must return within 30 days for evaluation.

INTERVENTIONS:
Dietary Supplement: Chlorella pyrenoidosa — Functional food, organically pressed into tablets (Registration with Anvisa/MS/Brazil: 6.7273.000)
  Arms: Experimental Group Chlorella pyrenoidosa (Outpatient phase)
Device: High Definition Transcranial Direct Current Stimulation — Neuromodulation Technics, non invasive, target and safety
  Other Names: HD-tDCS
  Arms: Experimental Group HD-tDCS (Hospital fase); Sham Group (Hospital Fase)

SUMMARY:
Reduced ejection fraction heart failure (HFrEF) is a complex and multifactorial condition. It is characterized by a decrease in the ability of the left ventricle to eject blood effectively during systole, resulting in an ejection fraction of less than 40%. This insufficiency in blood pumping leads to inadequate tissue perfusion and a series of adverse physiological adaptations that further compromise cardiac function, representing an important challenge in conducting treatment. The pathophysiology of HFrEF involves multiple mechanisms starting from the remodeling of the left ventricle in the face of some initial aggression, such as a heart attack, which culminates in a progressive deterioration of the contractile function. Additionally, neurohormonal systems are activated in response to the decrease in cardiac output, resulting in hyperactivation of the sympathetic nervous system and the renin-angiotensin-aldosterone axis, which leads to the activation of inflammatory cascades, mainly involving Interleukin 6 (IL-6) and Tumor Necrosis Factor Alpha (TNF-alfa), and disease progression. HFrEF is more prevalent in elderly populations and leads to increased hospital admissions. Furthermore, B12 depletion is more common in the elderly population and these two associated factors, functional impairment of the heart, disruption in the inflammatory cascade and depletion of nutrients, such as vitamin B12, can impact patients; quality of life in the long term. The reduction in B12 levels leads to changes in the cardiac and brain systems, due to the increase in homocysteine and the triggering of the inflammatory cascade. B12 supplementation through Chlorella Pyrenoidosa (microalgae - functional food) reduces cardiac damage and modulate the inflammatory cascade. And also High-Density Transcranial Direct Current Stimulation (HD-tDCS), a non-invasive technique capable of modulating neuronal excitability and inducing anti-inflammatory effects. In this sense, the objective is to evaluate the effects of HD-tDCS and the consumption of Chlorella Pyrenidosa to improve B12 levels and inflammatory response in patients with HFrEF.

DETAILED DESCRIPTION:
This study is a controlled, double-blind, randomized, crossover model clinical trial involving 28 participants with HFrEF admitted to a hospital for surgery and post-surgical outpatient care. Assessments will be carried out at baseline and after treatments through nutritional, clinical and laboratory assessment. The protocol is divided into two phases: the hospital phase with the implementation of the HD-tDCS protocol and the outpatient phase with the implementation of the Chlorella Pyrenoidosa protocol. The randomization of participants divides them into two groups: the active group that receives the intervention and the sham/control group that does not receive the intervention. In the hospital phase of the research, the protocol with HD-tDCS must be started before the surgical procedure, consisting of 5 sessions, applied once a day, for a period of up to 5 days before surgery, with stimulation in the Dorsolateral Prefrontal Cortex, with an intensity of 4mA and duration of 20 minutes each, with anodal stimulus. After post-surgery, at hospital discharge, the washout period of the groups is considered, in this phase another assessment of the group is considered and these are inverted, where the sham group in the previous phase becomes the active group at this stage and vice versa. The active group will receive the intervention through Chlorella pyreinodosa, the protocol in this phase is guided by the consumption of Chlorella p. in a home environment for 30 days until returning for evaluation from surgery, with the active group consuming 10 tablets, 5g/day, containing 4mcg of B12 from organic Chlorella pyrenoidosa in tablets (Registration with Health Surveillance (Anvisa)/Ministry of Health (MS)/Brazil No. 6.7273.000 - classification of functional food) during a period of thirty days and de control group will not receive. After this period, the active group and the control group must return for nutritional assessment and collection of final exams.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable HFrEF diagnosis and surgical indication;
* Adults and elderly people (20 to 80 years old);
* Able to respond to commands and give consent to participate in the research;
* Able to respond to simple commands and provide informed consent.

Exclusion Criteria:

* Patients with a clinical history of neuromuscular or cognitive instability,
* Pregnancy and contraindications for receiving neurostimulation (such as cardiac pacemakers and metallic brain implants);
* Patients with contraindications to the use of Chlorella (gastritis, esophagitis, peptic ulcers),;
* Patients with stroke and tumors.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Change B12 | After five days and after thirty days
  Change B12 (above 148pmol/L)
IL-6 Blood Analysis Biochemical | After five days and after thirty days
  Change IL-6 (below 10p/mL)
TNF alfa Blood Analysis Biochemical | After five days and after thirty days
  Change TNF alfa (below 2,8p/g/mL)

SECONDARY OUTCOMES:
Change Methylmalonic Acid Blood Analysis Biochemical | After five days and after thirty days
  Change Methylmalonic Acid (below 270nmol/L)
Change Homocysteine Blood Analysis Biochemical | After five days and after thirty days
  Change Homocysteine (below 12nmol/L)
Change Pro_BNP Blood Analysis Biochemical | After five days and after thirty days
  Change Pro_BNP (below 1000pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa M Cintra, Msc, Principal Investigator — Federal University of Paraiba
Locations (1):
- Federal University of Paraíba, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No